CLINICAL TRIAL: NCT01497119
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel Group Study of JNJ-39758979 in Adult Japanese Subjects With Moderate Atopic Dermatitis
Brief Title: A Study of JNJ-39758979 in Adult Japanese Patients With Moderate Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated prematurely due to 2 cases of agranulocytosis.
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR017455; 39758979ADM2001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Dermatitis, Atopic
Keywords: Moderate atopic dermatitis; JNJ-39758979; Japanese patients
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- JNJ-39758979, 300 mg (Experimental)
  Interventions: Drug: JNJ-39758979, 300 mg
- JNJ-39758979, 100 mg (Experimental)
  Interventions: Drug: JNJ-39758979, 100 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-39758979, 300 mg — Type=exact number, unit=mg, number=300, form=tablet, route=oral use, once daily for 6 weeks.
  Arms: JNJ-39758979, 300 mg
Drug: JNJ-39758979, 100 mg — Type=exact number, unit=mg, number=100, form=tablet, route=oral use, once daily for 6 weeks.
  Arms: JNJ-39758979, 100 mg
Drug: Placebo — Form=tablet, route=oral use, once daily for 6 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of JNJ-39758979 in adult Japanese patients with moderate, active atopic dermatitis.

DETAILED DESCRIPTION:
This is a randomized (treatment assigned by chance), double-blind (patient and investigator will not know what treatment is being given), multicenter, parallel-group, exploratory study in adult Japanese patients with moderate atopic dermatitis. This study will include 3 phases. In the screening phase, patients' eligibility will be determined. During the treatment phase, eligible patients will receive JNJ-39758979, 300 or 100 mg once daily, or placebo (a treatment that looks like JNJ-39758979, but contains no active agent) for up to 6 weeks. Study visits will occur at the end of Weeks 1, 2, 4, and 6. There will be a follow-up visit 4 weeks after dosing is complete. The duration of participation in the study for an individual patient may be up to 14 weeks (including screening). Patient safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of atopic dermatitis based on the criteria of the Japanese Dermatological Association and have: pruritus (itching); eczema-like changes in a typical pattern, and a chronic or chronically relapsing course.
* Childhood onset (under age of 13) of atopic dermatitis.
* Diagnosis of moderate atopic dermatitis based on the Rajka Langeland score between 4.5 and 7.5, inclusive.
* Have at least 3 ratings of "Moderate itching", "Severe itching", or "Extremely severe itching" either at night or during the day based on the Pruritus Categorical Response Scale (PCRS) in the 7 days prior to randomization.
* Atopic dermatitis with 10% to 50% (inclusive) Body Surface Area (BSA) involvement.

Exclusion Criteria:

* Have current signs or symptoms of liver or renal insufficiency or cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, psychiatric, or metabolic disturbances that are severe, progressive or uncontrolled in the Investigator's opinion. Patients with well controlled asthma, allergic rhinitis, or allergic conjunctivitis are allowed to participate. Atopic dermatitis patients with other chronic conditions will not be excluded if the Investigator has determined that the condition is not severe or progressive and is being controlled with stable therapy.
* Have any known malignancy or have a history of malignancy (with the exception of basal cell carcinoma, squamous cell carcinoma in situ of the skin, or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence within 5 years prior to the first administration of study agent).
* Evidence of any other skin condition that, in the opinion of the Investigator, would interfere with the assessment of atopic dermatitis.
* Use of non-steroid immunosuppressive or immunomodulatory agents within 4 weeks of randomization, including cyclosporine A, azathioprine, mycophenolate mofetil, and interferon gamma.
* Use of systemic corticosteroids within 4 weeks of randomization.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Monitoring of clinical laboratory tests | Up to approximately 14 weeks
  Assessments of blood, serum, and urine as a meaure of safety
The number of adverse events | Up to approximately 14 weeks
  As a measure of safety
Monitoring of electrocardiograms | Up to approximately 14 weeks
  As a measure of safety
Monitoring of vital signs tests | Up to approximately 14 weeks
  Blood pressure and pulse as a measure of safety
EASI (Eczema Area and Severity Index) score | Up to approximately 14 weeks
  A measure of the severity and extent of atopic dermatitis
Monitoring of physical examination assessments | Up to 10 weeks
  Including height and body weight, as a measure of safety

SECONDARY OUTCOMES:
Investigator's Global Assessment (IGA) | Up to approximately 14 weeks
  A 6-point scale that ranges from 0 (clear) to 5 (very severe disease).
Pruritus Categorical Response Scale (PCRS) | Up to approximately 14 weeks
  A 5-point categorical response scale where the response options range from "no itching" to "extremely severe itching."
Pruritus Numeric Rating Scales (PNRS) | Up to approximately 14 weeks
  An 11-point (0 to 10) numeric rating scale.
Pruritus Interference Numeric Rating Scale (PINRS) | Up to approximately 14 weeks
  An 11-point numerical rating scale of 0 to 10, where 0 = "Did Not Interfere" and 10 = "Completely Interfered."
Subject's Global Impressions of Change in Pruritus (SGICP) | Up to 10 weeks
  A 7-point scale ranging from "a lot more now" to " a lot less now" with a neutral center point ("neither more nor less").

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (13):
- Japan (13):
  - Chitose
  - Dazaifu
  - Ebetsu
  - Eniwa
  - Fukuoka
  - Kasuga
  - Matsudo
  - Saitama
  - Sapporo
  - Setagaya City
  - Tokyo
  - Utsunomiya
  - Yokohama